CLINICAL TRIAL: NCT07088198
Title: Joshi's Step With Buccal Mucosal Graft Urethroplasty in Nearly Obliterated Bulbar Urethral Stricture: A Prospective Study
Brief Title: Joshi's Step With Buccal Mucosal Graft Urethroplasty in Nearly Obliterated Bulbar Urethral Stricture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR661/4/24
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Joshi's Step; Buccal Mucosal Graft; Urethroplasty; Obliterated Bulbar Urethral Stricture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients will undergo dorsal onlay buccal mucosal graft urethroplasty with Joshi's step
  Interventions: Procedure: Joshi's step

INTERVENTIONS:
Procedure: Joshi's step — Patients will undergo dorsal onlay buccal mucosal graft urethroplasty with Joshi's step

SUMMARY:
This study aims to evaluate the functional and surgical outcome of Joshi's step with buccal graft urethroplasty for the management of nearly obliterated bulbar urethral stricture.

DETAILED DESCRIPTION:
Urethroplasty is a rapidly evolving art that continually improves and reinvents itself. After a century of silence, during which the anastomotic repair was the only solution for approaching the strictured urethra, the 1990s can be considered the Renaissance period for reconstructive urology.

In 2022, Joshi and Kulkarni introduced a new step to the augmented urethroplasty, particularly in patients with extremely narrow strictures where a single augmentation was insufficient. They avoid any resection of the residual native urethral plate, marking the narrowest portion. Then, the edges of the mucosa are reapproximated with interrupted suturing in a proper non-resecting approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary bulbar urethral stricture.
* Patients with non-traumatic bulbar urethral stricture.
* Patients with nearly obliterated bulbar urethral stricture, with the narrowest portion of the stricture is less than 1.5 cm in length.

Exclusion Criteria:

* Patients with traumatic bulbar urethral stricture.
* Patients with redo bulbar urethral stricture.
* Patients with obliterated bulbar urethral stricture.
* Patients with nearly obliterated long bulbar urethral stricture.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with primary bulbar urethral stricture
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 6 months postoperatively
  Incidence of success rate will be recorded.

SECONDARY OUTCOMES:
Urine flow rate | 6 months postoperatively
  Urine flow rate will be recorded.
The urethral lumen | 6 months postoperatively
  The urethral lumen by ascending urethrogram will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.